CLINICAL TRIAL: NCT05105061
Title: Intramuscular Ketamine Administration for the Treatment of Acute Suicidal Ideation With Concurrent EEG Monitoring
Brief Title: Intramuscular Ketamine for Suicidal Ideation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Matthew Klein, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY-20-01496; 21-1174 (Other: American Foundation for Suicide Prevention)
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Suicidal Ideation
Keywords: Suicide; EEG; Ketamine
MeSH Terms: conditions — Suicidal Ideation; Suicide | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine (1) then Placebo (2) (Experimental): Participants will receive an intramuscular injection of racemic ketamine, followed the next day by an intramuscular injection of saline (placebo)
  Interventions: Drug: Ketamine (Ketalar); Drug: Placebo
- Placebo (1) then Ketamine (2) (Placebo Comparator): Participants will receive an intramuscular injection of saline (placebo), followed the next day by an intramuscular injection of racemic ketamine
  Interventions: Drug: Ketamine (Ketalar); Drug: Placebo

INTERVENTIONS:
Drug: Ketamine (Ketalar) — 0.5 mg/kg of body weight
Drug: Placebo — IM injection of matching placebo

SUMMARY:
The objective of the present research protocol, a cross-over, subject-blinded, clinical trial, is to correlate changes in brain activity with reduction in suicidal ideation in response to a single intramuscular dose of ketamine. While ketamine is increasingly used as a rapid, antidepressant agent, there is accumulating evidence of additional anti-suicidal properties that may be distinct from its effects on depression. This pilot study will be used to determine (1) whether specific electroencephalogram (EEG) findings are correlated with response of SI to intramuscular (IM) ketamine, and (2) the effectiveness of IM ketamine in the treatment of acute SI.

ELIGIBILITY:
Inclusion Criteria:

* Current clinically significant suicidal ideation, defined as a score of > or = 4 on the MADRS item 10 and a positive answer on items 3,4 or 5 of the C-SSRS.
* Inpatient status at the time of study initiation.
* 18 to 70 years of age
* Capacity to consent

Exclusion criteria:

* Diagnosis of a primary psychotic disorder (e.g., schizoaffective disorder)
* Diagnosis of pervasive developmental disorder
* Diagnosis of a major neurocognitive disorder
* A positive urine pregnancy test
* Currently breastfeeding
* Drug or alcohol abuse or dependence within the preceding 3 months; a rather narrow time period was chosen, however, in order to allow participation by individuals with a history of substance abuse or dependence problems that could be secondary to their SI, and to more closely approximate patients seen in real-world settings. Given the increasingly widespread use of marijuana, and in an effort to recruit a naturalistic study population, concurrent marijuana use is not an exclusion criterion, as long as they are not actively intoxicated.
* Current positive UTOX for amphetamine, benzodiazepines, cocaine, opiates (if not prescribed)
* Medical issues or laboratory abnormalities requiring acute intervention
* Patients for whom an increase in blood pressure or intracranial pressure would pose a serious risk (e.g., aneurysmal vascular disease, arteriovenous malformation, history of intracerebral hemorrhage, unstable angina)
* Any lifetime history of ketamine or phencyclidine abuse
* A known hypersensitivity to or history of a serious adverse effect from to ketamine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Change in Auditory Mismatch Negativity (EEG) | Baseline and One hour post injection
  Change in Mismatch Negativity (MMN) amplitude or latency from baseline up to one hour after injection.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) #10 (SI) | Baseline and 24 hours post injection
  Change in MADRS #10 from baseline to 24 hours post-injection. Score range from 0-5, with higher score indicating higher severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Klein, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data will be made available the completion of the study.